CLINICAL TRIAL: NCT05831150
Title: Investigating Factors Affecting Clinical Trial Participation Rates in Patients With Esophageal Cancer
Brief Title: Discovering Patterns in Experiences of Patients in Esophageal Cancer Clinical Research
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 82828643
Record Dates: First submitted 2023-04-14; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Esophageal Cancer
Keywords: esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Participation in clinical trials usually favors a particular demographic group. But there is limited research available to explain what study attributes affect the completion of these specific demographic groups.

This study will investigate the safety and efficacy of esophageal cancer treatments. The focus will be on tracking the rates of completion and withdrawal among these individuals.

It will also try to analyze data from the perspective of different demographic groups to check for recurring trends which might yield insights for the sake of future esophageal cancer research.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age
* Diagnosis of esophageal cancer
* Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

* Women of childbearing potential without a negative pregnancy test; or women who are lactating.
* Has a serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Inability to perform regular electronic reporting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are actively considering involvement in an observational esophageal cancer clinical trial, but have not yet completed enrollment and registration.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to enroll in a clinical research. | 3 months
Number of study participants who remain in clinical research until completion. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kim HJ, Bains MS. Randomized clinical trials in esophageal cancer. Surg Oncol Clin N Am. 2002 Jan;11(1):89-109, viii. doi: 10.1016/s1055-3207(03)00076-0. PMID 11928803
- [Background] Harada K, Rogers JE, Iwatsuki M, Yamashita K, Baba H, Ajani JA. Recent advances in treating oesophageal cancer. F1000Res. 2020 Oct 1;9:F1000 Faculty Rev-1189. doi: 10.12688/f1000research.22926.1. eCollection 2020. PMID 33042518
- [Background] Zhou N, Hofstetter WL. Prognostic and therapeutic molecular markers in the clinical management of esophageal cancer. Expert Rev Mol Diagn. 2020 Apr;20(4):401-411. doi: 10.1080/14737159.2020.1731307. Epub 2020 Feb 24. PMID 32067548

DOCUMENTS (1):
  • Informed Consent Form (2023-04-13): https://cdn.clinicaltrials.gov/large-docs/50/NCT05831150/ICF_000.pdf